CLINICAL TRIAL: NCT05583682
Title: Clinical Performance of Nano-filled Resin-modified Glass Ionomer and Sub-micron Hybrid Resin Composite Restorations in Permanent Molar Teeth:18-month Randomised Clinical Trial
Brief Title: Clinical Performance of Resin-modified Glass Ionomer and Composite Restorations in Permanent Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacinlioglu, Nadya Marie (Other)
Collaborators: Yeditepe University (Other)
Responsible Party: Principal Investigator, Nadya Marie Hacinlioglu, Associate Professor, Cyprus Health and Social Sciences University, Hacinlioglu, Nadya Marie
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT1103200802
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Dental Caries in Children
Keywords: nano-filled resin-modified glass ionomer; sub-micron hybrid resin composite; permanent molar teeth

STUDY DESIGN:
Intervention Model Description: One of the Nano-filled glass ionomer or sub-micron hybrid resin composite restorative materials were applied to carious mandibular first molar teeth
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nano-filled resin-modified glass ionomer restoration (Experimental): One of the carious mandibular first molar teeth will be restored according to randomisation with nano-filled resin-modified glass ionomer restorative material (Ketac N 100/3M ESPE, USA)
  Interventions: Other: Dental restoration
- Sub-micron hybrid resin composite (Experimental): One of the carious mandibular first molar teeth will be restored according to randomisation with sub-micron hybrid resin composite restorative material (Spectrum TPH3, Dentsply Caulk, USA)
  Interventions: Other: Dental restoration

INTERVENTIONS:
Other: Dental restoration — Restoration of carious mandibular first molar teeth are restored either with nano-filled resin modified glass ionomer or sub-micron resin composite restorative material

SUMMARY:
The aim of this randomised controlled double-blinded, split mouth, single-center clinical trial was to evaluate the 18-month clinical performance of nano-filled resin-modified glass ionomer and sub-micron hybrid resin composite restorations in lower first permanent teeth of pediatric patients.

DETAILED DESCRIPTION:
Occlusal carious lesions on the left and right mandibular first molar teeth of 96 pediatric patients (54 female, 42 male) were restored in a split-mouth study design. Nano-filled resin-modified glass ionomer (Nano-RMGIC) (Ketac N 100, 3M/ESPE, USA) was used to restore the carious lesions for patients in the treatment group while a sub-micron hybrid resin composite (SpectrumTPH3, Dentsply, USA) was used for patients in the control group. Clinical evaluation of restorations were performed at the 1st week, 6th, 12th and 18th month recalls by two calibrated examiners according to the Modified-USPHS criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with two comparable occlusal carious lesions on both mandibular first permanent molars.
2. Neutral occlusion with a natural antagonist tooth
3. Patients that are able to come to recalls
4. Patients with a good oral hygiene

Exclusion Criteria:

1. Patients suffering systemic diseases or allergies
2. Patients with gastrointestinal problems
3. Mandibular first molar teeth with restorations
4. Patients with oral habits
5. Patients receiving orthodontic treatment
6. Hypomineralized or Hypoplastic first molars

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2008-05-01 (Actual); Primary Completion 2009-11-01 (Actual); Study Completion 2009-11-01 (Actual)

PRIMARY OUTCOMES:
Color Match | Changes of dental restorations regarding color match were observed at 1st week, 6th,12th and 18th month recalls.
  Color match of dental restorations were observed with a Vita Scale visually by two calibrated examiners. Restorations were scored Alfa, Bravo or Charlie according to Modified USPHS criteria. ( Alfa: Imperceptible in room light in one-second glance, Bravo: Perceptible mismatch with the Vita scale but clinically acceptable, Charlie: Esthetically unacceptable)
Marginal Discoloration | Changes of dental restorations regarding color match were observed at 1st week, 6th,12th and 18th month recalls.
  Marginal discoloration of dental restorations were observed by two calibrated examiners with visual inspection. Restorations were scored Alfa, Bravo or Charlie according to Modified USPHS criteria. (Alfa: No existing marginal discoloration, Bravo:Presence of discoloration at margins between restoration and tooth structure; discoloration does not penetrate towards the pulp, Charlie: The discoloration penetrated along the margins of the restoration in a pulpal direction.
Anatomic Form | Changes of dental restorations regarding color match were observed at 1st week, 6th,12th and 18th month recalls.
  Anatomic form of dental restorations were observed by two calibrated examiners by visual inspection and explorer. Restorations were scored Alfa, Bravo or Charlie according to Modified USPHS criteria. (Alfa: The restoration is not under-contoured, Bravo: The restoration is under-contoured, but there is no dentin or base exposed, Charlie: Sufficient restorative material is missing so that dentin or base is exposed.
Marginal Integrity | Changes of dental restorations regarding color match were observed at 1st week, 6th,12th and 18th month recalls.
  Marginal integrity of dental restorations were observed by two calibrated examiners with visual inspection and explorer. Restorations were scored Alfa, Bravo or Charlie according to Modified USPHS criteria. (Alfa: No visible evidence of a crevice along the margin into which an explorer will catch, Bravo: The explorer catches a crevice along the margin but there is no exposure of dentin or base, Charlie: Visible evidence of a crevice with exposure of dentin or base.)
Recurrent Decay | Changes of dental restorations regarding color match were observed at 1st week, 6th,12th and 18th month recalls.
  Recurrent decay of dental restorations were observed by two calibrated examiners with visual inspection. Restorations were scored Alfa or Charlie according to Modified USPHS criteria. (Alfa: No evidence of recurrent caries along the margin of the restoration, Charlie: Evidence of caries along the margin of the restoration.)
Fracture | Changes of dental restorations regarding color match were observed at 1st week, 6th,12th and 18th month recalls.
  Fracture of dental restorations were observed by two calibrated examiners by visual inspection with explorer. Restorations were scored Alfa, Bravo or Charlie according to Modified USPHS criteria. (Alfa: No fracture, Bravo: Small chip, but clinically acceptable, Charlie: Failure due to bulk restoration fracture.)
Surface Texture | Changes of dental restorations regarding color match were observed at 1st week, 6th,12th and 18th month recalls.
  Surface texture of dental restorations were observed by two calibrated examiners by visual inspection and explorer. Restorations were scored Alfa, Bravo or Charlie according to Modified USPHS criteria. (Alfa: Enamel like surface, Bravo: Surface rougher then enamel, clinically acceptable, Charlie: Surface unacceptable rough.)
Postoperative Sensitivity | Changes of dental restorations regarding color match were observed at 1st week, 6th,12th and 18th month recalls.
  Postoperative sensitivity of patients were assessed by two calibrated examiners by cold thermal test. Restorations were scored Alfa or Charlie according to Modified USPHS criteria. (Alfa: No sensitivity, Charlie: Sensitivity present.)

CONTACTS AND LOCATIONS:
Overall Officials: Nadya M Hacinlioglu-Ozpar, PhD, Principal Investigator — Cyprus Health and Social Sciences University

IPD SHARING:
Plan to Share IPD: No